CLINICAL TRIAL: NCT00000871
Title: A Phase II Safety and Immunogenicity Trial of Live Recombinant Canarypox ALVAC-HIV vCP205 With or Without HIV-1 SF-2 RGP120 in HIV-1 Uninfected Adult Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 202/HIVNET 014; HIVNET 014; 10589 (Registry Identifier: DAIDS ES Registry Number); AVEG 202
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; AIDS Vaccines; HIV Seronegativity; Avipoxvirus; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1
Biological: MN rgp120/HIV-1 and A244 rgp120/HIV-1
Biological: ALVAC-HIV MN120TMG (vCP205)
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To expand the available data regarding the safety and immunogenicity of 2 HIV-1 vaccine strategies: canarypox vector vCP205, or vCP205 with SF-2 rgp120. [AS PER AMENDMENT 7/2/98: To obtain immunogenicity and safety data on gp120 subunits that may induce enhanced neutralizing antibody response to primary isolates of HIV-1 in the context of previous immunization with a canarypox vector expressing HIV antigens (vCP205). To evaluate cytotoxic T lymphocyte responses at 1 and 2 years after initial vaccination with vCP205 plus rgp120 SF-2 or vCP205 alone.] In previous ALVAC vCP205/SF-2 rgp 120 studies, patients have developed antibodies that neutralize homologous laboratory strains; over 50% of patients have developed CD8+ cytotoxic T-lymphocyte responses to HIV env and gag epitopes at some point in the study. This Phase II study seeks to confirm these results among persons at lower or higher risk for HIV infection with a new lot of ALVAC vCP205, at a dose that is suitable for potential large-scale trials. [AS PER AMENDMENT 7/2/98: Addition of AIDSVAX B/B or AIDSVAX B/E boosts starting at least 12 months after receiving rgp120 or ALVAC vaccines may induce enhanced neutralizing antibody response as deemed from prior studies and thus is planned as "follow-up" therapy.]

DETAILED DESCRIPTION:
In previous ALVAC vCP205/SF-2 rgp 120 studies, patients have developed antibodies that neutralize homologous laboratory strains; over 50% of patients have developed CD8+ cytotoxic T-lymphocyte responses to HIV env and gag epitopes at some point in the study. This Phase II study seeks to confirm these results among persons at lower or higher risk for HIV infection with a new lot of ALVAC vCP205, at a dose that is suitable for potential large-scale trials. [AS PER AMENDMENT 7/2/98: Addition of AIDSVAX B/B or AIDSVAX B/E boosts starting at least 12 months after receiving rgp120 or ALVAC vaccines may induce enhanced neutralizing antibody response as deemed from prior studies and thus is planned as "follow-up" therapy.]

Volunteers are recruited and screened; those who are enrolled are then stratified by their risk status into 2 groups: individuals having lower-risk behavior for HIV and individuals having higher-risk behavior for HIV. Volunteers are then randomly assigned to arm A, B, or C and receive immunizations at months 0, 1, 3, and 6 as follows:

Group A- ALVAC vCP205 plus SF-2 rgp120 in MF59. Group B- ALVAC vCP205 plus saline placebo. Group C- Placebo-ALVAC plus saline placebo. [AS PER AMENDMENT 7/2/98: Beginning 12-18 months after initial vaccination, then 2, 6, and 12 months later, 10 volunteers from group A receive saline placebo, while 50 volunteers each from groups B and C are rerandomized within their respective groups, and are treated as follows.

Group B (subgroup 1) - AIDSVAX B/B. Group B (subgroup 2) - AIDSVAX B/E. Group B (subgroup 3) - alum placebo. Group C (subgroup 1) - AIDSVAX B/B. Group C (subgroup 2) - AIDSVAX B/E. Group C (subgroup 3) - alum placebo.] Volunteers are followed for 2 years and are tested for humoral immune response to HIV-1. Neutralizing activity to HIV-1 is performed on a subset of volunteers monitored for CTL response. [AS PER AMENDMENT 7/2/98: Volunteers receiving AIDSVAX B/B and AIDSVAX B/E will additionally be studied for formation of various neutralizing antibodies and parameters of cellular immunity.] [AS PER AMENDMENT 4/30/99: Because the subunit boosts that were added in version 3.0 are not available, the subunit boost portion of version 3.0 is cancelled.]

ELIGIBILITY:
Inclusion Criteria

Participants must have:

* Negative ELISA for HIV within 8 weeks of immunization.
* Normal history and physical examination.
* Availability for follow-up for planned duration of at least 24 months and willing to have 2 brief evaluations at 36 and 48 months.

Exclusion Criteria

Co-existing Condition:

Participants with the following symptoms or conditions are excluded:

* Active syphilis.

NOTE:

* AS PER AMENDMENT 6/25/97:
* Participant eligible if the serology is documented to be a false positive or due to adequately treated infection.
* Active tuberculosis (TB).

NOTE:

* Participant eligible if positive purified protein derivative and normal chest x-ray shows no evidence of TB and does not require isoniazid therapy.

Participants with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, malignancy, idiopathic anaphylaxis (AS PER AMENDMENT 6/25/97) or autoimmune disease. Participants with a history of cancer are excluded unless they have undergone surgery followed by a sufficient observation period to give a reasonable assurance of cure.
* Any history of anaphylaxis or history of other serious adverse reactions to vaccines.
* Immediate-type hypersensitivity reaction to egg products or neomycin (used to prepare ALVAC vaccines).

Prior Medication:

Excluded:

* Immunosuppressive medications.
* Live attenuated vaccines within 60 days of study.
* Use of investigational agents within 30 days prior to study.
* Prior receipt of HIV-1 vaccines or placebo recipient in a previous HIV vaccine trial.

Prior Treatment:

Excluded:

* Receipt of blood products or immunoglobulin within past 6 months.

Risk Behavior:

Excluded:

* Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol. Specifically excluded are persons with a history of suicide attempts within 3 years, recent suicidal ideation or who have past or present psychosis.
* Medically indicated subunit or killed vaccines, e.g., influenza, pneumococcal, hepatitis A and B allowed provided administered more than 2 weeks from HIV study immunizations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420
Dates: Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belshe R, Study Chair; Gorse G, Study Chair
Locations (18):
- United States (18):
  - UAB AVEG, Birmingham, Alabama
  - Public Health Enterprises Foundation, Inc. HIVNET, San Francisco, California
  - Denver Dept. of Health HIVNET, Denver, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Cook County Hospital HIVNET, Chicago, Illinois
  - Univ. of Illinois at Chicago HIVNET, Chicago, Illinois
  - JHU AVEG, Baltimore, Maryland
  - Fenway Community Health Center HIVNET, Boston, Massachusetts
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - NY Blood Ctr. HIVNET, New York, New York
  - NY Univ. Med. Ctr. HIVNET, New York, New York
  - Univ. of Rochester AVEG, Rochester, New York
  - Univ. of Pennsylvania HIVNET, Philadelphia, Pennsylvania
  - Memorial Hosp. of Rhode Island HIVNET, Providence, Rhode Island
  - The Miriam Hosp. HIVNET, Providence, Rhode Island
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington
  - Uw Hivnet, Seattle, Washington

REFERENCES:
- [Background] Belshe RB, Stevens C, Gorse G, Buchbinder S, Sridhara R, Self S, Weinhold K, Sheppard H, Duliege AM, Meignier B, McNamara J, Flores J (NIAID AVEG, HIVNET Vaccine Development Groups). Phase II evaluation of a live recombinant canarypox (ALVAC) vector HIV-1 vaccine with or without gp120 subunit HIV-1 vaccine. 13th Meeting, International Society for Sexually Transmitted Diseases Research, 1999 Jul 11-14 [227].
- [Background] Gorse GJ, Patel GB, Mandava MD, Arbuckle JA, Doyle TM, Belshe RB; National Institute of Allergy and Infectious Diseases AIDS Vaccine Evaluation Group. Cytokine responses to human immunodeficiency virus type 1 (HIV-1) induced by immunization with live recombinant canarypox virus vaccine expressing HIV-1 genes boosted by HIV-1(SF-2) recombinant GP120. Vaccine. 2001 Feb 8;19(13-14):1806-19. doi: 10.1016/s0264-410x(00)00378-9. PMID 11166906
- [Background] Belshe RB, Stevens C, Gorse GJ, Buchbinder S, Weinhold K, Sheppard H, Stablein D, Self S, McNamara J, Frey S, Flores J, Excler JL, Klein M, Habib RE, Duliege AM, Harro C, Corey L, Keefer M, Mulligan M, Wright P, Celum C, Judson F, Mayer K, McKirnan D, Marmor M, Woody G; National Institute of Allergy and Infectious Diseases AIDS Vaccine Evaluation Group and HIV Network for Prevention Trials (HIVNET). Safety and immunogenicity of a canarypox-vectored human immunodeficiency virus Type 1 vaccine with or without gp120: a phase 2 study in higher- and lower-risk volunteers. J Infect Dis. 2001 May 1;183(9):1343-52. doi: 10.1086/319863. Epub 2001 Apr 10. PMID 11294665
- [Background] Worku S, Gorse GJ, Belshe RB, Hoft DF. Canarypox vaccines induce antigen-specific human gammadelta T cells capable of interferon-gamma production. J Infect Dis. 2001 Sep 1;184(5):525-32. doi: 10.1086/322792. Epub 2001 Jul 26. PMID 11474428
- [Background] Gorse GJ, Patel GB, Belshe RB; National Institute of Allergy and Infectious Diseases HIV Vaccine Trials Network. HIV type 1 vaccine-induced T cell memory and cytotoxic T lymphocyte responses in HIV type 1-uninfected volunteers. AIDS Res Hum Retroviruses. 2001 Aug 10;17(12):1175-89. doi: 10.1089/088922201316912781. PMID 11522187